CLINICAL TRIAL: NCT04575506
Title: Influence of the Diversity and Composition of the Microbiota in the Development of Pediatric Fatty Liver: Identification of Biomarkers and Development of Personalized Therapy: The MicroKid Project
Brief Title: Influence of the Diversity and Composition of the Microbiota in the Development of Pediatric Fatty Liver
Acronym: MicroKid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pública de Navarra (Other)
Collaborators: Complejo Hospitalario de Navarra (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI_2020/29
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2020-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity; Metabolic Syndrome
Keywords: Non-alcoholic hepatic steatosis; Obesity; Children; Exercise; Diet; Microbiota
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention)
- Obesity-Non-hepatic steatosis (Active Comparator): Healthy lifestyle education program focused on dietary and lifestyle guidelines for both children and parents (2 days/month, 60 min), and exercise program based on high-intensity interval training which combine aerobic and resistance training (at least 3 days/week, from 38 to 44 min).
  Interventions: Other: Multidisciplinary intervention program
- Obesity-Hepatic steatosis (Experimental): Healthy lifestyle education program focused on dietary and lifestyle guidelines for both children and parents (2 days/month, 60 min), and exercise program based on high-intensity interval training which combine aerobic and resistance training (at least 3 days/week, from 38 to 44 min).
  Interventions: Other: Multidisciplinary intervention program

INTERVENTIONS:
Other: Multidisciplinary intervention program — The intervention program includes an educational program promoting healthy dietary habits and physical activity (nutritionist and exercise physiologist) (2 times/month, for children and parents), and supervised home-based exercise (from 3 to 5 times/week, 38-44 min) program for 12-weeks.
  Arms: Obesity-Hepatic steatosis; Obesity-Non-hepatic steatosis

SUMMARY:
The objectives of the present study are: 1) to identify the intestinal and salivary microbiota associated with the presence and severity of hepatic steatosis in children (Study I: case-control study), and 2) to develop a personalized 12-week intervention program based on diet and exercise to examine its effects on the diversity and composition of the microbiota in children with hepatic steatosis (Study II: intervention study)

DETAILED DESCRIPTION:
The MicroKid project will acts first as a case-control study (Study I) in order to identify the hepatic steatosis and intestinal and salivary microbiota in children grouped as non-overweight, obese-non-hepatic steatosis, and obese-hepatic steatosis. Then, an intervention study (Study II) will be developed for those children with obesity (i.e., obese-non-hepatic steatosis, and obese-hepatic steatosis groups).

Methodology: A total of 60 children, 8-12 years-old, will be assigned to control (non-overweight children, N= 20), obese-non-hepatic steatosis (children with obesity, but without hepatic steatosis, N=20), and obese-hepatic steatosis (children with obesity and hepatic steatosis, N= 20) groups (Study I: case-control study). The obesity and obesity + hepatic steatosis groups will attend to a 12-weeks healthy lifestyle education program (2 days/month) and home-based exercise program (minimum 3 days/week) (Study II: intervention study).

The combined intervention program for the Study II will include: i) healthy lifestyle education program focused on dietary and lifestyle guidelines for both children and parents (2 days/month, 60 min), and ii) exercise program based on high-intensity interval training which combines aerobic and resistance training (at least 3 days/week, from 38 to 44 min).

Measurements: In the Study I (i.e., case-control study), all participants will be evaluated at baseline. For the Study II (i.e., intervention study), only those participants that belongs to obese-non-hepatic steatosis and obese-hepatic steatosis groups, will be additionally evaluated after the intervention program (12-week). The following outcomes will be measured: hepatic fat fraction and abdominal adiposity (magnetic resonance imaging), intestinal and salivary microbiota, body composition (bioimpedance), cardiometabolic risk factors, liver enzymes, physical fitness (field-fitness tests), physical activity (accelerometry), sleep (accelerometry), dietary habits (24h recalls, and food frequency questionnaires), and pubertal development and sociodemographic characteristics will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Obesity defined based on the sex-and-age specific body mass index standards
* 8-12 years old

Exclusion Criteria:

* Medical conditions that hamper their participation in the exercise program

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Hepatic fat | baseline and post-test (12-weeks)
  Hepatic fat fraction measured by magnetic resonance imaging before and after 12-weeks intervention program
Intestinal microbiota | baseline and post-test (12-weeks)
  Diversity and composition of intestinal microbiota before and after 12-weeks intervention program
Salivary microbiota | baseline and post-test (12-weeks)
  Diversity and composition of salivary microbiota before and after 12-weeks intervention program

SECONDARY OUTCOMES:
Visceral adiposity | baseline and post-test (12-weeks)
  Visceral adipose tissue measured by magnetic resonance imaging before and after 12-weeks intervention program
Subcutaneous abdominal adiposity | baseline and post-test (12-weeks)
  Subcutaneous abdominal adipose tissue measured by magnetic resonance imaging before and after 12-weeks intervention program
Intermuscular abdominal adiposity | baseline and post-test (12-weeks)
  Intermuscular abdominal adipose tissue measured by magnetic resonance imaging before and after 12-weeks intervention program
Weight | baseline and post-test (12-weeks)
  Weight measured by bioimpedance before and after 12-weeks intervention program
Height | baseline and post-test (12-weeks)
  Height measured by stadiometer before and after 12-weeks intervention program
Fat mass | baseline and post-test (12-weeks)
  Fat mass measured by bioimpedance before and after 12-weeks intervention program
Fat-free mass | baseline and post-test (12-weeks)
  Fat free mass measured by bioimpedance before and after 12-weeks intervention program
Glucose | baseline and post-test (12-weeks)
  Glucose measured by blood analysis before and after 12-weeks intervention program
Insulin | baseline and post-test (12-weeks)
  Serum insulin concentration measured by ELISA before and after 12-weeks intervention program
Cholesterol | baseline and post-test (12-weeks)
  Serum cholesterol measured by spectrophotometry before and after 12-weeks intervention program
Triglycerides | baseline and post-test (12-weeks)
  Serum triglycerides measured by spectrophotometry before and after 12-weeks intervention program
Leptin | baseline and post-test (12-weeks)
  Plasma leptin concentration measured by ELISA before and after 12-weeks intervention program
Adiponectin | baseline and post-test (12-weeks)
  Plasma adiponectin measured by ELISA before and after 12-weeks intervention program
C-reactive protein | baseline and post-test (12-weeks)
  Plasma hs-CRP measured by ELISA before and after 12-weeks intervention program
Waist circumference | baseline and post-test (12-weeks)
  Waist circumference measured by non-elastic tape before and after 12-weeks intervention program
Systolic and diastolic blood pressure | baseline and post-test (12-weeks)
  Systolic and diastolic blood pressure measured by sphygmomanometer before and after 12-weeks intervention program
Physical fitness | baseline and post-test (12-weeks)
  Cardiorespiratory fitness, upper- and lower-limbs, and speed agility measured by the Alpha-fitness battery.
Physical activity and sleep | baseline and post-test (12-weeks)
  Physical activity and sleep measured by accelerometry before and after 12-weeks intervention program
24h dietary habits | baseline and post-test (12-weeks)
  24h dietary habits assessed by 24h recalls before and after 12-weeks intervention program
Dietary habits history | baseline and post-test (12-weeks)
  Dietary habits history assessed by food frequency questionnaires before and after 12-weeks intervention program

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Complejo Hospitalario de Navarra, Pamplona
  - Public University of Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No